CLINICAL TRIAL: NCT02090023
Title: Long Term Prognosis of Taiwanese Patients With Obstructive Sleep Apnea
Brief Title: Long Term Prognosis of Taiwanese Patients With OSA
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 201309084RIND
Record Dates: First submitted 2014-03-16; First posted 2014-03-18 (Estimated); Last update posted 2014-03-18 (Estimated); Status verified 2014-03

CONDITIONS: Obstructive Sleep Apnea
Keywords: Obstructive sleep apnea; National Health Insurance Research Database in Taiwan; Survival Analysis; Validation Studies; Cohort Studies
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- NHIRD obstructive sleep apnea: Secondary database from community-based National Health Insurance Research Database
- NTUH obstructive sleep apnea cohort: Primary database from enrollment of retrospective NTUH hospital-based cohort

SUMMARY:
The purpose of this study is to explore long-term prognosis and to identify the predictors in Taiwanese OSA patients. Validation of the prediction model derived from NHIRD with the database of National Taiwan University Hospital (NTUH) sleep center is planed to determine the effects of different treatments on long-term prognosis.

DETAILED DESCRIPTION:
Obstructive sleep apnea (OSA) is a common disorder characterized by intermittent hypoxia and sleep fragmentation. OSA is associated with cardiovascular morbidity and mortality, metabolic dysregulation, and neurocognitive dysfunction, which may bring worse prognosis. Continuous positive airway pressure (CPAP) is the standard treatment of OSA while the oral appliance and surgery are the alternative treatments. The differences of craniofacial features among races contributed to the race-specific presentations of OSA. Up to date, only limited studies investigated the long-term prognosis of OSA and most of them recruited Caucasians and African Americans. Moreover, most studies didn't address the impact of treatment other than CPAP on the long-term prognosis. .

National Health Insurance Research Database (NHIRD) in Taiwan enrolled 99% of whole Taiwan's population and has longer period of 10 years for follow-up, which is suitable for investigation of long-term prognosis and predictors in OSA. However, due to limited parameters for diagnosis and treatment, the results could be biased in such secondary database research. Center of Sleep Disorder in National Taiwan University Hospital (NTUH) established from 2006 has 2,600 sleep studies annually. Therefore, database and cohort from sleep center could offer the validations of the prognosis and predictors determined from NHIRD. In addition, the impact of all three treatment modalities, namely CPAP, oral appliance, and surgery, on long-term prognosis could be studied in the prospective way.

Therefore, in this project, we aimed to achieve three goals (1) To explore long-term prognosis and identify the predictors in Taiwanese OSA patients with NHIRD, where the prediction mode of prognosis was established (2). To validate the prediction model derived from NHIRD with the database of NTUH sleep center (3) To determine the effects of different treatments on long-term prognosis with prospective following NTUH sleep center cohort.

ELIGIBILITY:
Inclusion Criteria:

* NHIRD - >=20 y/o; OSA ICD-9-CM code: 780.51,780.53,780.57, or 327.23; coexisted with PSG procedure code: 17008B,17008A.
* NTUH cohort - >=20 y/o; PSG AHI>5

Exclusion Criteria:

* patients refusing to anticipate our study

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Obstructive sleep apnea (PSG apnea-hypopnea index (AHI)>5 or The International Classification of Diseases, 9th Revision, Clinical Modification (ICD-9-CM) code:780.51,780.53,780.57, or 327.23) Community-based from NHIRD cohort Hospital-based from NTUH cohort
Sampling Method: Probability Sample
Enrollment: 4000 (Estimated)
Dates: Start 2014-01; Primary Completion 2017-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Death or Major adverse cardiovascular events(MACEs) | from 2000 to 2013, up to 13 years
  MACEs includes cardiogenic death, ischemic stroke, myocardial injury or acute coronary syndrome requiring revascularization.
  Data from NHIRD (database screening retrospectively) and NTUH cohort (recallable history taking).

SECONDARY OUTCOMES:
Cardiovascular morbidity | from 2000 to 2013, up to 13 years
  Timing and events of new onset of hypertension, atrial fibrillation, or atrial flutter
Neurocognitive morbidity, up to 13 years | from 2000 to 2013, up to 13 years
  Timing and events of traffic accident, new onset of depression, or dementia, or epilepsy.
Metabolic morbidity | from 2000 to 2013, up to 13 years
  Timing and events of incident diabetics or diabetic complications or new onset of dyslipidemia.
Other morbidity | from 2000 to 2013, up to 13 years
  Incidence of malignancy or chronic kidney disease.

CONTACTS AND LOCATIONS:
Overall Officials: Peilin Lee, Ph.D., Principal Investigator — National Taiwan University Hospital, Center of Sleep Disorders
Locations (1):
- Center of Sleep Disorder, Taipei, Taiwan